CLINICAL TRIAL: NCT04732338
Title: The Effectiveness of Osteopathic Manipulative Medicine in the Management of Headaches Associated With Post Concussion Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00001814
Record Dates: First submitted 2021-01-11; First posted 2021-02-01 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Headache; Post-Concussion Syndrome
MeSH Terms: conditions — Headache; Post-Concussion Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm - Osteopathic Manipulative Therapy (Experimental): Standard of care including physical therapy, occupational therapy and over the counter medication AND OMT as described below:
  1. Musculoskeletal examination of the cervical spine. Testing will be comprised of :
     1. Range of motion testing involving cervical rotation, lateral side bending, flexion and extension.
     2. Muscular palpation of the cervical paraspinals for hypertonicity of the muscles and/or tenderness.
  2. Patient placed supine on the examination table.
  3. Treatment sessions lasting 5-10 minutes each. OMT techniques: cervical muscle energy, myofascial release of the cervical paraspinals and a suboccipital release.
  Assessment with Headache Impact Test (HIT-6) at baseline and follow-up visit and change in pain scores between baseline and post treatment.
  Interventions: Other: Osteopathic Manipulative Therapy
- Control - Standard of care (No Intervention): Standard of care including physical therapy, occupational therapy and over the counter medication.

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy — Osteopathic Manipulative Therapy (OMT) is a non-pharmacological, noninvasive form of manual medicine. Osteopathic practitioners use a wide variety of therapeutic manual techniques to improve physiological function and help restore homeostasis in the body. There is a structural assessment is to identify possible abnormalities of tissue texture. Areas of asymmetry and misalignment of bony landmarks are also evaluated, along with the quality of motion, balance, and organization. These asymmetries, also known as somatic dysfunctions, are then treated by a variety of manual treatments, administered by osteopaths.
  Arms: Study arm - Osteopathic Manipulative Therapy

SUMMARY:
Pilot study looking at the Osteopathic Manipulative Treatment (OMT) for various headache types in patients with post-concussion syndrome (PCS). Twenty-six subjects with symptoms lasting >3 months were enrolled and were randomly assigned to a treatment group (n = 13) and a control group (n = 13).

DETAILED DESCRIPTION:
Evidence shows the effectiveness of Osteopathic Manipulative Treatment (OMT) for various headache types, with limited evidence of its use for headaches related to mild traumatic brain injury (MTBI). No studies were found regarding OMT for headaches in patients with post-concussion syndrome (PCS), defined as symptom persistence >3 months after MTBI.

Objective: To evaluate OMT for headaches in patients with PCS. Methods: A controlled pilot study was conducted of patients with PCS who presented to an outpatient interdisciplinary rehabilitation clinic. Twenty-six subjects with symptoms lasting >3 months were enrolled and were randomly assigned to a treatment group (n = 13) and a control group (n = 13). Primary outcome measures were 1) immediate change in headache scores with a visual analog scale (VAS) and 2) change in the 6-item Headache Impact Test (HIT-6) between baseline and follow-up visits. 10 control participants completed HIT-6 between baseline and follow-up visits but did not receive OMT and did not complete VAS. After OMT, immediate VAS changes in treatment group and the improvements in HIT-6 scores for both groups between baseline and follow-up were analyzed for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild traumatic brain injury (MTBI),
* age 18 years or older
* injury occurring >3 months prior, and
* headache as a primary symptomatic concern.

Exclusion Criteria:

* history of moderate to severe traumatic brain injury (TBI),
* documented intracranial injury,
* chronic headache or migraine headache before the injury,
* treatment with a headache specialist at the time of injury, or receipt of IV infusion for medication for headache at the time of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alphonsa Thomas, DO, Principal Investigator — HMH-JFK
Locations (1):
- Hackensack Meridian Health - JFK Medical Center, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. McCrory, P. Consensus Statement on Concussion in Sport, 3 rd International Conference on Concussion in Sport. Clinical Journal of Sport Medicine 2010, 20(4), 332. 2. Ellis, M. J.; Leddy, J. J.; Willer, B. Physiological, vestibule-ocular and cervicogenic post-concussion disorders: An evidence-based classification system with directions for treatment.Brain Injury 2014, 29(2), 238-248. 3. Langlois, J. A.; Rutland-Brown, W.; Wald, M. M. The epidemiology and impact of traumatic brain injury: a brief overview. Journal of Head Trauma Rehabilitation2006, 21(5), 375-378. 4. Willer, B.; Leddy, J. J. Management of Concussion and Post-Concussion Syndrome. Current Treatment Options in Neurology2006, 8(5), 415-426. 5. Anderson, T.; Heitger, M.; Macleod, A. D. Concussion and mild head injury. Practical Neurology2006, 6(6), 342-357. 6. Kushner, D. Mild Traumatic brain injury: toward understanding manifestations and treatment. Archives of Internal Medicine1998, 158(15), 1617. 7. Alexander, M. P. Mild traumatic brain injury: pathophysiology, natural history, and clinical management. Neurology1995, 45(7), 1253-1260. 8. Zasler, N. D., Katz, D. I., & Zafonte, R. D. (2007). Brain injury medicine: Principles and practice. New York: Demos 9. Hiploylee, C.; Dufort, P. A.; Davis, H. S.; Wennberg, R. A.; Tartaglia, M. C.; Mikulis, D.; Hazrati, L.-N.; Tator, C. H. Longitudinal Study of Postconcussion Syndrome: Not Everyone Recovers. Journal of Neurotrauma2017, 34(8), 1511-1523. 10. Cerritelli, Francesco et al. "Osteopathy for Primary Headache Patients: A Systematic Review." Journal of Pain Research 10 (2017): 601-611. PMC. Web. 20 Dec. 2017. 11. Espi-lopez, G.V, et al. "Do Manual Therapy techniques have a positive effect on quality of life in people with tension-type headache? A randomized controlled trial." European Journal of Physical Medicine and Rehabilitation2016, 52(4), 447-56. 12. Cerritelli, Francesco et al. "Osteopathy for Primary Headache Patients: A Systematic Review." Journal of Pain Research 2017: (15)601-611. PMC. Web. 20 Dec. 2017. 13. Castillo, I.; Wolf, K; Rakowsky, A. "Concussions and Osteopathic Manipulative Treatment: An Adolescent Case Presentation." J Am Osteopath Assoc 2016;116(3):178-181. doi: 10.7556/jaoa.2016.034. 14. Guernsey, D.; Leder, A.; Yao, S. "Resolution of Concussion Symptoms After Osteopathic Manipulative Treatment: A Case Report." J Am Osteopath Assoc 2016;116(3):e13-e17. doi: 10.7556/jaoa.2016.036. 15. Adragna et al. "Osteopathic manipulative treatment of headache in a polytrauma patient: case report." The Journal of Headache and Pain 2015, 16(Suppl 1):A181. 16. Savarese, R. G., Capobianco, J. D., & Cox, J. J., (2009). OMT Review 3rd edition.

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm - Osteopathic Manipulative Therapy: Standard of care including physical therapy, occupational therapy and over the counter medication AND OMT as described below:
  1. Musculoskeletal examination of the cervical spine. Testing will be comprised of :
     1. Range of motion testing involving cervical rotation, lateral side bending, flexion and extension.
     2. Muscular palpation of the cervical paraspinals for hypertonicity of the muscles and/or tenderness.
  2. Patient placed supine on the examination table.
  3. Treatment sessions lasting 5-10 minutes each. OMT techniques: cervical muscle energy, myofascial release of the cervical paraspinals and a suboccipital release.
  Assessment with Headache Impact Test (HIT-6) at baseline and follow-up visit and change in pain scores between baseline and post treatment.
  Osteopathic Manipulative Therapy: Osteopathic Manipulative Therapy (OMT) is a non-pharmacological, noninvasive form of manual medicine. Osteopathic practitioners use a wide variety of therapeutic manual techniques to improve physiological function and help restore homeostasis in the body. There is a structural assessment is to identify possible abnormalities of tissue texture. Areas of asymmetry and misalignment of bony landmarks are also evaluated, along with the quality of motion, balance, and organization. These asymmetries, also known as somatic dysfunctions, are then treated by a variety of manual treatments, administered by osteopaths.
Period: Overall Study
Arm/Group | Study Arm - Osteopathic Manipulative Therapy | Control - Standard of Care
Started | 13 | 13
Completed | 10 | 10
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm - Osteopathic Manipulative Therapy | Control - Standard of Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15) | 42 (17) | 43.5 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Immediate Change in Headache Scores With a Visual Analog Scale (VAS)
Description: Change in the headache scores, defined as the different pain pre and post treatment using the visual analog scale (VAS).
  VAS is widely used to capture pain, the scale ranges from 0-10 with 0 (best outcome) being no pain and 10 being the worst pain possible (worst outcome).
Time Frame: Same day with treatment on visit 1
Population: We captured the pre and post VAS score and the change between the two.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Arm - Osteopathic Manipulative Therapy | Control - Standard of Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Initial VAS score | 5.6 (1.7) | NA (NA) — VAS was not measured in the control group
  Post intervention VAS score | 3.5 (2.1) | NA (NA) — VAS was not measured in the control group
  Change in VAS score | 2 (1.8) | NA (NA) — VAS was not measured in the control group

2. Primary Outcome: Change in the 6-item Headache Impact Test (HIT-6) Between Baseline and Follow-up Visit.
Description: HIT-6 was completed at baseline and competed to HIT-6 completed post treatment at follow up visit.
  Headache Impact Test (HIT-6) is a measure of headache severity and provides information regarding the effect of headache on other domains related to functional participation. The HIT-6 has six questions and the range goes from 36 (best outcome) to a maximum score of 78 (worst outcome). Higher HIT-6 scores indicate increased headache severity and greater functional limitations.
Time Frame: 4 weeks post treatment (Follow-up visit 1)
Population: Pre and post intervention HIT-6 scores and change between the two.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Study Arm - Osteopathic Manipulative Therapy | Control - Standard of Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Initial HIT-6 score | 63.0 [57.8 to 70.0] | 62.0 [49.5 to 65.5]
  Post-intervention HIT-6 score | 60.0 [55.0 to 65.0] | 60.5 [49.5 to 64.3]
  Change in HIT-6 score | 3.5 [0.8 to 7.3] | 2.0 [-2.5 to 3.5]

ADVERSE EVENTS:
Time Frame: up to 6 weeks of post-treatment follow up
Arm/Group | Study Arm - Osteopathic Manipulative Therapy | Control - Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
We lost 3 patients in each group to follow-up as they did not come back although our team attempted to reach out to them.

Limitation: no VAS was measured in the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04732338/Prot_SAP_000.pdf